CLINICAL TRIAL: NCT02504840
Title: Thematic Studies of Multiple Sclerosis and Related Diseases
Brief Title: Natural History of Multiple Sclerosis and Its Mimickers
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150158; 15-N-0158
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Neurologic Disorders; Healthy Volunteers; Multiple Sclerosis
Keywords: Multiple Sclerosis; Clinically Isolated Syndrome; CNS Inflammatory Demyelination; Radiologically Isolated Syndrome; Natural History
MeSH Terms: conditions — Nervous System Diseases; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers: healthy volunteers
- patient controls: Participants with diseases that share features with MS.
- patients with suspected or confirmed multiple sclerosis: Participants with definite, probable, or possible MS.

SUMMARY:
Background:

- Magnetic resonance imaging (MRI) has been used for decades to help diagnose and monitor neurological disorders like multiple sclerosis (MS). Researchers want to improve how MRI pictures are taken. They also want to learn more about using newer MRIs with stronger magnets to get better pictures than standard MRIs provide.

Objectives:

- To collect data that will help researchers better understand MS and related diseases.

Eligibility:

* Adults 18 and older with MS or MRI findings that appear similar to MS, or with other neurological diseases that may look or act like MS.
* Healthy adult volunteers.

Design:

* Participants will be screened with a review of their medical records.
* Participants will have a baseline visit. It will include a physical exam, medical history, and neurological exam. They may have blood tests.
* The study will last indefinitely.
* Participants may have MRIs. Some MRIs may include a contrast dye. For this, a needle will be used to guide a thin plastic tube into an arm vein.
* Participants may have up to 2 lumbar punctures per year. Skin will be numbed and a needle inserted between back bones will remove fluid.
* Participants may give saliva samples and have an eye exam.
* Participants may have evoked potential tests. These measure how the nervous system responds to different types of stimulation. Participants may sit in front of a TV and watch pictures on the screen. Or they may wear earphones that make a clicking noise or static. Or they may get a small electrical shock that may tingle and cause a hand or foot twitch.
* Participants may have tests of strength, spasticity, sensations, balance, and/or walking.

DETAILED DESCRIPTION:
Objectives.

The goals of this protocol are to study the pathophysiology of multiple sclerosis (MS), primarily through small studies that utilize magnetic resonance imaging (MRI), and to correlate the results with clinical and biological measures. The protocol includes only techniques with minimal risk (standard and quantitative clinical evaluation, MRI, blood draws, saliva testing, urine and stool collection, visual evoked potentials, ophthalmologic evaluation) or more-than-minimal risk (injection of approved gadolinium-based contrast agents, lumbar punctures) that are appropriate and common in this study population. Under this protocol, we will conduct:

* Pilot substudies. These studies are exploratory and hypothesis generating. Once sufficient data are collected to justify a hypothesis-driven study and a formal power analysis, further work will continue under either a dedicated protocol or, if appropriate, a hypothesis-testing substudy. There are no enrollment limitations for pilot substudies.
* Hypothesis-testing substudy. These studies have a specific hypothesis that can be tested with at most 6 participants per arm. If additional participants are required, a memo will be sent to the Protocol Review Committee (PIRC) and its statistical reviewer to request review of a hypothesis-testing substudy for possible additional enrollment.The memo will also be forwarded to the IRB.
* Individual patient substudies. These studies seek to increase knowledge of a disease process or to assist in the diagnosis of an individual patient.
* Technique development substudies. These studies will lay the groundwork for new experimental paradigms, using the methods approved under this protocol, which can be further tested in the substudies listed above.
* Training of investigators. These studies will be done to train new investigators in techniques relevant to the studies under this protocol.

Study Population

Three groups of study participants will be enrolled:

* MS patients. Participants with definite, probable, or possible MS.
* Patient controls. Participants with diseases that share features with MS.
* Healthy volunteers.

Design

We will design small substudies as ideas arise in the course of our work that are pertinent to the theme of the pathophysiology of MS (or of diseases that share features with MS). If a hypothesis testing sub-study leads to results of interest and if a larger population is necessary to reach statistical significance, a separate protocol will be submitted with a priori hypotheses, specific study design and power analysis adapted from the pilot or exploratory substudies performed in the present protocol.

Outcome Measures

These will include MRI, clinical, and biological outcome measures consistent with the objectives of the study and its investigators. Imaging measures will focus on features related to the central nervous system (CNS), particularly focal lesions. Clinical measures will include standard and established MS disability scales as well as quantitative measures related to function. Biological measures will include genotype, gene expression, proteomics, virological studies, and immunological profiling.

ELIGIBILITY:
* INCLUSION CRITERIA:

<TAB>

* One or more of the following:

  * Diagnosis of MS, clinically isolated syndrome, or radiologically isolated syndrome.
  * Presentation with clinical or neuroimaging findings that, in the best judgment of the investigators, are possibly consistent with central nervous system inflammatory demyelination.
  * Healthy volunteer.
* Age greater than or equal to18.
* Able to participate in study procedures and provide high-quality clinical research data, in the best judgment of the investigators.
* Interest of the study investigators in performing one or more procedures under one or more of the substudies.

EXCLUSION CRITERIA:

<TAB>

* Unwilling to allow sharing and/or use in future studies of coded samples and data that are collected for this study.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 1300 participants will be enrolled onto this open-ended thematic protocol. The following study populations will be included:- Participants with definite, probable, or possible MS. These participants either carry a diagnosis of MS, or else their referring clinicians are considering the diagnosis.-Participants with diseases that share imaging features with MS. These participants report clinical symptoms or prior MRI findings that could, in the best judgment of the investigators, be due to inflammatory demyelination of the central nervous system.- Healthy volunteers.-Withdrawals and dropouts will not be replaced.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Association between clinical status and research data | over time
  Imaging measures will focus on features related to the central nervous system (CNS), particularly focal lesions. Clinical measures will include standard and established MS disability scales as well as quantitative measures related to function. Biological measures will include genotype, gene expression, proteomics, virological studies, and immunological profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gaitan MI, Shea CD, Evangelou IE, Stone RD, Fenton KM, Bielekova B, Massacesi L, Reich DS. Evolution of the blood-brain barrier in newly forming multiple sclerosis lesions. Ann Neurol. 2011 Jul;70(1):22-9. doi: 10.1002/ana.22472. Epub 2011 Jun 27. PMID 21710622
- [Background] Jones BC, Nair G, Shea CD, Crainiceanu CM, Cortese IC, Reich DS. Quantification of multiple-sclerosis-related brain atrophy in two heterogeneous MRI datasets using mixed-effects modeling. Neuroimage Clin. 2013 Aug 13;3:171-9. doi: 10.1016/j.nicl.2013.08.001. eCollection 2013. PMID 24179861
- [Background] McFarland HF, Frank JA, Albert PS, Smith ME, Martin R, Harris JO, Patronas N, Maloni H, McFarlin DE. Using gadolinium-enhanced magnetic resonance imaging lesions to monitor disease activity in multiple sclerosis. Ann Neurol. 1992 Dec;32(6):758-66. doi: 10.1002/ana.410320609. PMID 1471866
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-N-0158.html